CLINICAL TRIAL: NCT02563574
Title: Alcohol and HIV: Biobehavioral Interactions and Intervention
Brief Title: ARCH II Study (Alcohol Research Center on HIV Study II)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Brown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB201500625-N; 2P01AA019072-06 (NIH); OCR16162 (Other: Universiy of Florida)
Record Dates: First submitted 2015-09-28; First posted 2015-09-30 (Estimated); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Alcohol Consumption; HIV; Motivation
Keywords: Alcohol and brain function; HIV and brain function; Motivational Interviewing
MeSH Terms: conditions — Alcohol Drinking | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational Interviewing Group (Experimental): This group of participants will receive the motivational interviewing. In addition to blood specimen collection, a questionnaire assessment and neurocognitive assessments will also be performed.
  Interventions: Behavioral: Motivational Interviewing; Other: Questionnaire assessment; Other: Neurocognitive assessments; Other: Blood specimens
- Control Group (Active Comparator): This group of participants will not receive motivational interviewing. They will have blood specimen collection, questionnaire assessment, and neurocognitive assessments performed.
  Interventions: Other: Questionnaire assessment; Other: Neurocognitive assessments; Other: Blood specimens

INTERVENTIONS:
Behavioral: Motivational Interviewing — A type of counseling aimed at reducing consumption of alcohol.
  Arms: Motivational Interviewing Group
Other: Questionnaire assessment — Several different types of questionnaires will be fill out by the participants.
Other: Neurocognitive assessments — Several different types of neurocognitive assessment will be performed.
Other: Blood specimens — Blood specimens will be used to measure the immunological, virologic, and hepatic status, as well as other biomarkers.

SUMMARY:
This study is being done to learn about the interaction of alcohol consumption and HIV on brain function. The proposed study will have two broad objectives. The first is to incorporate functional neuroimaging (FMRI) approaches, along with additional Magnetic Resonance Spectroscopy (MRS) methods that will enable a delineation in both functional and cerebral metabolic disturbances affecting specific functional brain systems that are associated with the interaction of ethanol (ETOH) consumption on Human Immunodeficiency Virus (HIV)-associated brain dysfunction. Recent data indicate that HIV infected patients with heavy ETOH consumption have FMRI abnormalities and exhibit alterations on other neuroimaging measures compared to moderate drinkers and people who do not drink at all. The second objective is to examine the extent to which reductions in ETOH consumption among heavy drinkers with HIV infection result from a motivational intervention. The findings from this study will provide important information on how heavy ETOH and HIV interact to affect the brain functional responsiveness, and the extent of improvement that might be gained by reducing heavy ETOH use.

DETAILED DESCRIPTION:
In this research study, participants will be randomized (much like flipping a coin) by a computer program to either no counseling or FMRI during the baseline visit in the second session for this visit.

Each time point (baseline, 3 months and 9 months) consists of 2 participant sessions. Session 1) at baseline is for the purposes of recruiting and determining if participants meet study criteria; during all visits, study criteria are reviewed to ensure that enrolled participants are still eligible. After determining eligibility, study information is explained by the research assistant and consent is then obtained. Additional psychiatric and substance use assessment and neurological and will be performed. Blood and urine specimens will be obtained and sent to lab for measurement of immunological, virologic, and hepatic status and other biomarkers. The remainder of the blood specimens will be frozen and banked for future analyses. All blood specimens banks for future analyses will be deidentified. A neurocognitive assessment performed by a research assistant. The duration will be approximately 120 minutes. Session 2) will occur within one week of visit one. It will consist of an MRI scan lasting approximately 50 minutes. Functional imaging will be conducted during this MRI time. All participants will undergo all procedures at baseline, and three and nine months.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected;
* English speaking;
* Physically mobile;
* Willingness to participate in the Motivational Interviewing (MI) to reduce ETOH consumption.

Exclusion Criteria:

* Neurological disorders;
* Evidence of dementia;
* Past opportunistic brain infection;
* Major psychiatric illness;
* Current major psychiatric disturbance;
* Unstable medical conditions (cancer);
* MRI contraindications (e.g., pregnancy, claustrophobia, metal implants);
* Physical impairment precluding motor response or lying still.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-12; Primary Completion 2021-12-16 (Actual); Study Completion 2021-12-16 (Actual)

PRIMARY OUTCOMES:
FMRI images will be performed for changes in the brain between the groups | Baseline and 6 month follow-up
  Cerebral metabolite abnormalities

SECONDARY OUTCOMES:
Structured Clinical Interview for Diagnostic and Statistical Manual (DSM)-IV (SCID) | Baseline
  A structured interview given to participants in order to assess current and past alcohol use and dependence
Lifetime Alcohol and Drug Use History | Baseline
  This interview will be conducted at baseline to gather information about age of onset of alcohol use, period of heaviest drinking, most drinks consumed on a single day, and number of drug classes used lifetime.
Kreek-McHugh-Schluger-Kellogg (KMSK) Scale | Baseline, 3-month, 6-month, and 12-month follow-ups.
  Developed as a research measure of drug use severity in accordance with DSM-IV criteria, the KMSK is reliable and valid, quantifying frequency, duration, and amount of individual drug use.
Timeline Followback (TLFB) | Baseline, 3-month, 6-month, and 12-month follow-ups.
  The TLFB interview will be used to assess recent alcohol use at baseline, as well as during the follow-up intervals. The TLFB interview is a calendar-assisted structured interview which provides a way to cue memory so that accurate recall is enhanced. The TLFB will provide data on the percentage of drinking days, drinks consumed per week, and the percentage of heavy drinking days.
Urine Drug Screen | Baseline, 3-month, 6-month, and 12-month follow-ups.
  Urine drug screens will be performed using Varian's TestCup Pro5, testing for benzodiazepines, amphetamines, opiates, & cocaine.
Short Inventory of Problems (SIP) | Baseline, 3-month, 6-month, and 12-month follow-ups.
  The SIP assesses 15 negative consequences of alcohol use over the chosen time period (in this case 3 months) and has been found to have good psychometric properties. Maximum score is 45
Epworth Sleepiness Scale (ESS) | Baseline, 3-month, 6-month, and 12-month follow-ups.
  The ESS proposes eight daytime scenarios, and the participant is asked to rate how likely they are to fall asleep in each situation on a four-point scale (0-3).
Center for Epidemiological Studies-Depression Scale (CES-D) | Baseline, 3-month, 6-month, and 12-month follow-ups.
  A 20-item screening test for depression and depressive disorder
Beck Anxiety Inventory | Baseline, 3-month, 6-month, and 12-month follow-ups.
  21-question multiple-choice self-report inventory that is used for measuring the severity of anxiety
Early Life Stress Questionnaire (ELSQ) | Baseline
  A 5-section self-report questionnaire assessment of adverse childhood events
The Frontal System Behavioral Scale (FrSBe) | Baseline, 3-month, 6-month, and 12-month follow-ups.
  A 46-item self-report questionnaire designed to measure behavior related to frontal systems damage
Medical Outcomes Study HIV Health Survey (MOS-HIV) | Baseline, 3-month, 6-month, and 12-month follow-ups.
  A 35-item self-report questionnaire designed in order to assess functional status and well-being among HIV-positive individuals
Montreal Cognitive Assessment (MoCA) | Baseline, 3-month, 6-month, and 12-month follow-ups.
  measurement used to screen for dementia and mild cognitive impairment
Hopkins Verelan Learning Test Revised (HVLT-R) | Baseline, 3-month, 6-month, and 12-month follow-ups.
  cognitive assessment that measures verbal learning and memory
Brief Visuospatial Memory Test Revised (BVMT-R) | Baseline, 3-month, 6-month, and 12-month follow-ups.
  A measure of visuospatial memory
Paced Auditory Serial Addition Test (PASAT-1) | Baseline, 3-month, 6-month, and 12-month follow-ups.
  A cognitive assessment which measures visuospatial memory
WAIS-3 Letter Number Sequencing | Baseline, 3-month, 6-month, and 12-month follow-ups.
  7-item cognitive assessment with a total of 21 maximum points
WAIS-3 Digit Symbol | Baseline, 3-month, 6-month, and 12-month follow-ups.
  A timed neuropsychological test sensitive to brain damage, dementia, age and depression consisting of digit-symbol pairs followed by a list of digits
WAIS-3 Symbol Search | Baseline, 3-month, 6-month, and 12-month follow-ups.
  Cognitive assessment measuring processing speed with a total max score of
Trail Making | Baseline, 3-month, 6-month, and 12-month follow-ups.
  timed cognitive assessment looking at working memory and executive functioning
Grooved Pegboard | Baseline, 3-month, 6-month, and 12-month follow-ups.
  measures performance speed in a fine motor task
Stroop Task | Baseline, 3-month, 6-month, and 12-month follow-ups.
  timed cognitive task
Verbal Fluency | Baseline, 3-month, 6-month, and 12-month follow-ups.
  timed language measure
Animal Fluency | Baseline, 3-month, 6-month, and 12-month follow-ups.
  timed language measure
The Wechsler Test of Adult Reading (WTAR) | Baseline, 3-month, 6-month, and 12-month follow-ups.
  cognitive tast measuring verbal intelligence
Boston Naming Test | Baseline, 3-month, 6-month, and 12-month follow-ups.
Adaptive Rate Continuous Performance Test (ARCPT) | Baseline, 3-month, 6-month, and 12-month follow-ups.
  computerized adaptive task measuring attention
California Computerized Assessment Package (CalCAP) | Baseline, 3-month, 6-month, and 12-month follow-ups.
  computerized task measuring reaction time

CONTACTS AND LOCATIONS:
Overall Officials: Ron Cohen, Ph.D, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - University of Florida, Gainesville, Florida
  - Florida International University, Miami, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Scott K, Guy AA, Zelaya DG, Surace A, Elwy AR, Keuroghlian AS, Mayer KH, Monti PM, Kahler CW. Research and engagement considerations for alcohol use telehealth services within HIV care: a qualitative exploration in federally qualified health centers. AIDS Care. 2023 Nov;35(11):1786-1795. doi: 10.1080/09540121.2023.2197640. Epub 2023 Apr 11. PMID 37039068